CLINICAL TRIAL: NCT06346314
Title: Is There an Immediate Effect on Pectoralis Minor Length After Performing a Prone Scapular Retraction Exercise Using Typical Sets and Repetitions in Pain Free Participants
Brief Title: Is There an Immediate Effect on Pectoralis Minor Length After Performing a Prone Scapular Retraction Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrews University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12241976
Record Dates: First submitted 2024-02-28; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2023-11

CONDITIONS: Pectoralis Minor Length
Keywords: Pectoralis Minor; Reciprocal Inhibition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Participants who underwent intervention.
  Interventions: Other: Scapular retraction exercise

INTERVENTIONS:
Other: Scapular retraction exercise — Participant lies prone with hands superior to the head on a treatment plinth and lifts their elbows 10 repetitions for three sets with 30 seconds of rest between each set.

SUMMARY:
The goal of this clinical trial is to test normal participants.

The main question it aims to answer is:

• Do the participant's pectoralis minor muscles change length immediately after performing an exercise that recruits the scapular retractor muscles? Participants will have their pectoralis minor muscle measured, then perform an exercise recruiting the scapular retractor muscles, and then have their pectoralis muscle measured again.

DETAILED DESCRIPTION:
The participants will have their standing height measured in centimeters with a tape measure fixed against a wall. Participants will then step away from the wall and will be asked to stand in their normal resting position. A mark will be placed on the most medial-inferior aspect of the coracoid process and a second mark on the anterior-inferior edge of the third rib, one index finger's width lateral to the sternum. A caliper will then be used to measure the distance between these marks as the participant holds a normal exhalation.

Participants will then lay prone on a treatment plinth with a small towel roll under their forehead. The participants will form both fists and place them on the plinth just superior to their head, with bilateral thumbs up and the ulnar side of the hands resting on the plinth, and their arms relaxed so their elbows remain on the plinth. The participants will then lift their elbows off the plinth as high as possible while keeping their hands on the plinth. The participants will repeat this motion for 10 repetitions, performing three sets of this exercise with 30 seconds of rest in between each set.

After the third set, the participants will stand up and a second caliper will be used to once again measure PM length by the same tester using the same marks. This will conclude the testing procedure and the participant's involvement in the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older. At least 130 degrees of shoulder elevation. None of the exclusion criteria.

Exclusion Criteria:

* Current shoulder pathology and or pain, prior shoulder surgery, any neurological impairment, any upper quarter deformity, a fracture of the upper extremity, or systemic inflammatory disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Pectoralis Minor Length | Measured before and immediately after intervention
  Length of the Pectoralis Muscle length in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Dye, MPT, Principal Investigator — North Idaho Physical Therapy
Locations (1):
- North Idaho Physical Therapy, Hayden, Idaho, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borstad JD. Measurement of pectoralis minor muscle length: validation and clinical application. J Orthop Sports Phys Ther. 2008 Apr;38(4):169-74. doi: 10.2519/jospt.2008.2723. Epub 2007 Nov 21. PMID 18434665
- [Background] Viriyatharakij N, Chinkulprasert C, Rakthim N, Patumrat J, Ketruang B. Change of pectoralis minor length, and acromial distance, during scapular retraction at 60 degrees shoulder elevation. J Bodyw Mov Ther. 2017 Jan;21(1):53-57. doi: 10.1016/j.jbmt.2016.04.015. Epub 2016 Apr 29. PMID 28167190

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT06346314/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT06346314/ICF_001.pdf